CLINICAL TRIAL: NCT07385092
Title: The Effect of Continuous Monitoring Versus Routine Spot-checks on Altered Vital Signs in Patients Recovering From Non-cardiac Surgery on Normal Wards: the "COME ON, NOW!" Trial
Brief Title: Continuous Vital Sign Monitoring Versus Routine Spot-checks in Patients After Non-cardiac Surgery
Acronym: COME ON NOW
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Kristen Thomsen, MD, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-101178-BO-ff
Record Dates: First submitted 2026-01-13; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Vital Sign Monitoring; Post Operative Complications; Non-cardiac Surgery; RCT; Anesthesiology
Keywords: continuous vital signs; vital signs; vital sign monitoring; post-operative care; anesthesiology; anesthesia; hypotension; post-operative complications
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will be blinded to group allocation. Clinicians and investigators will be blinded to continuous vital signs in the control group. In the intervention group, clinicians will receive information on vital signs from the study staff. Data analysts are blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blinded continuous vital sign monitoring (Sham Comparator): Continuous ward monitoring with vital signs recorded but not available to patients, clinicians, or investigators.
  Interventions: Device: Blinded continuous vital sign monitoring
- Unblinded continuous vital sign monitoring (Experimental): Continuous ward monitoring with vital signs available to investigators.
  Interventions: Device: Unblinded continuous vital sign monitoring

INTERVENTIONS:
Device: Unblinded continuous vital sign monitoring — Continuous ward monitoring with vital signs available to investigators. Oxygen saturation, blood pressure (intermittent in intervals of 60 minutes), heart rate, and respiratory rate will be continuously measured and streamed to the investigators (specifically, to a central monitor). The investigators will alert nurses or physicians when SpO2 is <85% for ≥2 minutes, respiratory rate is <7/min or >30/min for ≥2 minutes, MAP is <60 mmHg, or heart rate is <45 bpm or >130 bpm for ≥2 minutes, or in case of apnea for ≥1 minute - supplemented by clinical judgement and the complete electronic record. Investigators will alert clinicians when concerning patterns are identified, whether or not alerts have been triggered. Clinicians will determine if response is necessary and what interventions might be appropriate.
  Arms: Unblinded continuous vital sign monitoring
Device: Blinded continuous vital sign monitoring — Continuous ward monitoring with vital signs recorded but not available to patients, clinicians, or investigators.
  Arms: Blinded continuous vital sign monitoring

SUMMARY:
The "COME ON, NOW!" trial is a randomized, single-center trial in patients recovering from non-cardiac surgery on normal wards investigating whether continuous vital sign monitoring - compared to routine spot-checks by nurses - reduces the total duration of abnormal vital signs per hour during the first 48 hours after admission to the normal ward.

DETAILED DESCRIPTION:
"Surgery went well, and everything is fine. Your relative is still in the operating room, but you can visit her/him this afternoon on the normal ward." Each day, thousands of patient families receive relieving calls like this. A call better reflecting clinical reality would be: "Surgery went well, and everything is fine so far - but the most dangerous time is still ahead. The postoperative period poses a much higher risk for patients than surgery itself." Indeed, rates of major postoperative complications and death remain frighteningly high. If the month after surgery were considered a disease, it would be the third leading cause of death worldwide. Most major complications and deaths occur during the initial hospitalization, under direct medical care.

Postoperative deterioration is usually preceded by changes in vital signs minutes to hours earlier. However, these alterations are frequently missed because vital signs on normal wards are typically assessed only every 4-8 hours. Continuous monitoring may allow earlier detection of instability and enable timely interventions to prevent or mitigate serious complications.

The investgators therefore propose a single-center randomized trial in adults recovering from major non-cardiac surgery on normal wards to compare continuous postoperative vital sign monitoring with routine intermittent spot-checks. Patients will be randomized to blinded or unblinded continuous monitoring using a wearable, wireless sensor system (Radius VSM, Masimo, Irvine, CA). In the unblinded group, clinicians will receive real-time alerts.

The primary outcome will be the cumulative duration of vital sign abnormalities during the first 48 hours on the ward. Secondary outcomes will include clinical interventions triggered by these abnormalities. Exploratorily, the investigators will assess a composite of serious in-hospital complications.

Our long-term goal is to reduce postoperative morbidity and mortality by enabling earlier recognition of clinical deterioration and timely intervention on general wards.

ELIGIBILITY:
Inclusion Criteria:

Consenting patients ≥45 years scheduled for elective abdominal surgery with planned postoperative admission to a normal ward after an overnight stay in an advanced post-anesthesia care unit.

Exclusion Criteria:

* Emergency surgery
* Pregnancy
* Impossibility to perform continuous monitoring with the Radius VSM sensor (Masimo, Irvine, CA)
* Atrial fibrillation
* Patients designated Do Not Resuscitate, or are receiving end-of-life care

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Total duration of abnormal vital signs | 48 hours after admission to the normal ward
  Total duration of abnormal vital signs per hour (minutes per hour) during the first 48 hours after admission to the normal ward, i.e., the minutes per hour patients have any of the following abnormal vital signs ("any versus none"): peripheral oxygen saturation (SpO2) <85%, mean arterial pressure (MAP) <60 mmHg, heart rate <45 bpm or >130 bpm, and respiratory rate <7/min or >30/min.

SECONDARY OUTCOMES:
Individual components of the composite primary endpoint | 48 hours after admission to the normal ward
  Total duration of a SpO2 <85% per hour (minutes per hour)
Individual components of the composite primary endpoint | 48 hours after admission to the normal ward
  Total duration of a MAP <60 mmHg per hour (minutes per hour)
Individual components of the composite primary endpoint | 48 hours after admission to the normal ward
  Total duration of a heart rate <45 bpm per hour (minutes per hour)
Individual components of the composite primary endpoint | 48 hours after admission to the normal ward
  Total duration of a heart rate >130 bpm per hour (minutes per hour)
Individual components of the composite primary endpoint | 48 hours after admission to the normal ward
  Total duration of a respiratory rate <7/min per hour (minutes per hour)
Individual components of the composite primary endpoint | 48 hours after admission to the normal ward
  Total duration of a respiratory rate >30/min per hour (minutes per hour)
Quantitative metrics of peripheral oxygen saturation | 48 hours after admission to the normal ward
  Area under a SpO2 of 85% (SpO2 <85% x min)
Quantitative metrics of peripheral oxygen saturation | 48 hours after admission to the normal ward
  Time-weighted average hypoxemia (SpO2 <85% x min / total monitoring time)
Quantitative metrics of peripheral oxygen saturation | 48 hours after admission to the normal ward
  Number of SpO2 <85% events per patient
Quantitative metrics of peripheral oxygen saturation | 48 hours after admission to the normal ward
  Proportion of patients with any SpO2 <85% event
Quantitative metrics of peripheral oxygen saturation | 48 hours after admission to the normal ward
  Total cumulative duration of SpO2 <85%
Quantitative metrics of mean arterial pressure | 48 hours after admission to the normal ward
  Area under a MAP of 60 mmHg (mmHg x min)
Quantitative metrics of mean arterial pressure | 48 hours after admission to the normal ward
  Time-weighted average hypotension (MAP <60 mmHg x min / total monitoring time)
Quantitative metrics of mean arterial pressure | 48 hours after admission to the normal ward
  Number of MAP <60 mmHg events per patient
Quantitative metrics of mean arterial pressure | 48 hours after admission to the normal ward
  Proportion of patients with any MAP <60 mmHg event
Quantitative metrics of mean arterial pressure | 48 hours after admission to the normal ward
  Total cumulative duration of MAP <60 mmHg
Quantitative metrics of heart rate | 48 hours after admission to the normal ward
  Area under a heart rate of 45 bpm (<45 bpm x min)
Quantitative metrics of heart rate | 48 hours after admission to the normal ward
  Area above a heart rate of 130 bpm (>130 bpm x min)
Quantitative metrics of heart rate | 48 hours after admission to the normal ward
  Time-weighted average bradycardia (<45 bpm x min / total monitoring time)
Quantitative metrics of heart rate | 48 hours after admission to the normal ward
  Time-weighted average tachycardia (>130 bpm x min / total monitoring time)
Quantitative metrics of heart rate | 48 hours after admission to the normal ward
  Number of events per patient with heart rate <45 bpm
Quantitative metrics of heart rate | 48 hours after admission to the normal ward
  Number of events per patient with heart rate >130 bpm
Quantitative metrics of heart rate | 48 hours after admission to the normal ward
  Proportion of patients with any event with heart rate <45 bpm
Quantitative metrics of heart rate | 48 hours after admission to the normal ward
  Proportion of patients with any event with heart rate >130 bpm
Quantitative metrics of heart rate | 48 hours after admission to the normal ward
  Total cumulative duration of heart rate <45 bpm
Quantitative metrics of heart rate | 48 hours after admission to the normal ward
  Total cumulative duration of heart rate >130 bpm
Quantitative metrics of respiratory rate | 48 hours after admission to the normal ward
  Area under a respiratory rate 7/min (<7/min x min)
Quantitative metrics of respiratory rate | 48 hours after admission to the normal ward
  Area above a respiratory rate 30/min (>30/min x min)
Quantitative metrics of respiratory rate | 48 hours after admission to the normal ward
  Time-weighted average bradypnea (<7/min x min / total monitoring time)
Quantitative metrics of respiratory rate | 48 hours after admission to the normal ward
  Time-weighted average tachypnea (>30/min x min / total monitoring time)
Quantitative metrics of respiratory rate | 48 hours after admission to the normal ward
  Number of events per patient with respiratory rate <7/min
Quantitative metrics of respiratory rate | 48 hours after admission to the normal ward
  Number of events per patient with respiratory rate >30/min
Quantitative metrics of respiratory rate | 48 hours after admission to the normal ward
  Proportion of patients with any event with respiratory rate <7/min
Quantitative metrics of respiratory rate | 48 hours after admission to the normal ward
  Proportion of patients with any event with respiratory rate >30/min
Quantitative metrics of respiratory rate | 48 hours after admission to the normal ward
  Total cumulative duration of respiratory rate <7/min
Quantitative metrics of respiratory rate | 48 hours after admission to the normal ward
  Total cumulative duration of respiratory rate >30/min
The incidence of a composite of clinical interventions for desaturation, hypoventilation, tachypnea, tachycardia, bradycardia, and hypotension. | 48 hours after admission to the normal ward
  Clinical responses will be considered interventions if:
  1. they are documented in the medical record, and
  2. meet at least one of the following criteria:
     * Respiratory treatment if preceded within 2 hours by SpO2 <85% or respiratory rate <7/min and investigator alert: oxygen, inhaled bronchodilators, naloxone, diuretics, and ventilatory support.
     * Tachycardia interventions preceded within 2 hours by a heart rate of >130 bpm and investigator alert, excluding chronically used preoperative medications: beta-blockers, calcium channel blockers, amiodarone, adenosine, and cardioversion.
     * Bradycardia interventions preceded within 2 hours by a heart rate <45 bpm and investigator alert: Isoproterenol, atropine, glycopyrrolate, epinephrine, cardiac pacing, cardioversion.
     * Hypotension interventions preceded within 2 hours by a mean arterial pressure <60 mmHg and investigator alerts: crystalloids, colloids, norepinephrine, albumin.
     * Any activation of the rapid response team or ICU transfer.

OTHER OUTCOMES:
Composite of serious in-hospital complications | 48 hours after admission to the normal ward
  The investigators will also record components of our exploratory composite of serious in-hospital complications, including naloxone administration, rapid-response team activation, unplanned ICU transfer, revision surgery, infectious complications, myocardial infarction, stroke, unplanned tracheal intubation, non-fatal cardiac arrest, and death during the first 48 hours after admission to the normal ward and during hospital stay.
Time-to-event endpoint | 30 days after index surgery
  Time-to-event endpoint with the event "hospital discharge" within 30 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Saugel, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No